CLINICAL TRIAL: NCT00140322
Title: Dane County Safety Assessment for Elders (SAFE) Research Study
Brief Title: Dane County Safety Assessment (SAFE) Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Wisconsin Department of Health and Family Services (Other Government); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3954; U17/CCU522465
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Falls
Keywords: falls; injury; elderly
MeSH Terms: conditions — Wounds and Injuries | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise, fall risk reduction

SUMMARY:
A randomized controlled trial to assess the effectiveness of an at-home comprehensive approach to preventing falls among adults 65 years and older at high risk for falls.

DETAILED DESCRIPTION:
A randomized controlled trial to assess the effectiveness of a comprehensive approach to preventing falls among adults 65 years and older at high risk for falls. This intervention includes a comprehensive health assessment in each participant's home combined with tailored risk reduction strategies such as individualized strength and balance exercises. The study is also conducting a community-based program to engage and educate physicians about fall prevention.

The goal of the study is to demonstrate a 40% decrease in fall rates. Other expected outcomes include decreased hospital and nursing home stays, improved physical function, and a decreased fear of falling.

ELIGIBILITY:
Inclusion Criteria: Adults age 65+, at high risk for falls, -

Exclusion Criteria: Adults <65 years

-

Ages: 0 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 455
Dates: Start 2002-10; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Decreased fall rates

SECONDARY OUTCOMES:
decreased hospital and nursing home stays
improved physical function
decreased fear of falling

CONTACTS AND LOCATIONS:
Overall Officials: Jane Mahoney, MD, Principal Investigator — University of Wisconsin Medical School

REFERENCES:
- [Derived] Garbez N, Mbatchi LC, Maseda E, Luque S, Grau S, Wallis SC, Muller L, Lipman J, Roberts JA, Lefrant JY, Roger C. A Loading Micafungin Dose in Critically Ill Patients Undergoing Continuous Venovenous Hemofiltration or Continuous Venovenous Hemodiafiltration: A Population Pharmacokinetic Analysis. Ther Drug Monit. 2021 Dec 1;43(6):747-755. doi: 10.1097/FTD.0000000000000874. PMID 33560097